CLINICAL TRIAL: NCT00685776
Title: A 76-Week, Worldwide, Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Assess the Tolerability and Efficacy of Anacetrapib When Added to Ongoing Therapy With a Statin in Patients With Coronary Heart Disease (CHD) or CHD Risk-Equivalent Disease
Brief Title: Study to Assess the Tolerability and Efficacy of Anacetrapib in Patients With Coronary Heart Disease (CHD) or CHD Risk-Equivalent Disease (MK-0859-019)
Acronym: DEFINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0859-019; 2007_648 (Other: Merck Study Number)
Record Dates: First submitted 2008-05-23; First posted 2008-05-28 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Coronary Heart Disease (CHD); CHD Risk-Equivalent Disease
Keywords: CHD/CHD risk-equivalent disease; Coronary Heart Disease (CHD)
MeSH Terms: conditions — Coronary Disease | interventions — anacetrapib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anacetrapib (Experimental): Participants randomly assigned to anacetrapib in base study will continue same treatment if enrolled in study extension.
  Interventions: Drug: anacetrapib
- Placebo (Placebo Comparator): Participants randomly assigned to placebo in base study will continue same treatment if enrolled in study extension.
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: anacetrapib — Participants will receive one tablet of anacetrapib 100 mg once daily for 76 weeks.
  Other Names: MK0859
  Arms: Anacetrapib
Drug: Comparator: placebo — Participants will receive one placebo tablet once daily for 76 weeks.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy of anacetrapib (100 mg) for 24 weeks relative to placebo, on plasma concentrations of Low Density Lipoprotein Cholesterol and assess the safety and tolerability of anacetrapib (100 mg) in participants with CHD/CHD risk-equivalent disease on stable dose regimen of statin with or without other lipid-modifying therapy. The two year extension to this study will further evaluate the long-term safety profile and efficacy of anacetrapib in CHD/CHD-risk equivalent patients who are on ongoing therapy with a statin with or without other lipid-modifying therapy.

DETAILED DESCRIPTION:
The 76 week treatment period is followed by a 12 week reversibility phase which can be extended by up to another 12 weeks in order to allow participants who have completed their week 88 visit to continue in the study until the Extension study is ready to be implemented.

In the optional extension, participants will be assigned to the same treatment arm to which they were assigned in the base study. The total duration of the extension study will be up to 116 weeks; which will include a 2 year treatment period, followed by a 12 week reversal phase. A post-extension study follow-up phone call will be completed 12 weeks after discontinuation or completion of study treatment. Participants previously treated with anacetrapib or placebo will be invited in a 4:1 ratio in an optional extended reversal phase. The total duration of the extended reversal phase will be 1 year.

Participants previously treated with anacetrapib in the DEFINE study will be followed periodically for up to 4 years to determine plasma levels of anacetrapib. Participants will also be invited to participate in a sub-study consisting of one clinic visit to measure anacetrapib levels in the plasma and the subcutaneous adipose tissue.

ACRONYM: DEFINE= Determining the EFficacy and Tolerability of Cholesteryl ester transfer protein (CETP) INhibition with AnacEtrapib

ELIGIBILITY:
Inclusion Criteria:

* Base Study:

  * Patient has Coronary Heart Disease (CHD) or CHD Risk-Equivalent Disease and is treated with a statin, with well controlled LDL-C
* Extension Study:

  * Patient has completed the base study including the reversibility period (i.e. 12 or to up to 24 weeks).
  * Patient is on statin therapy ± lipid-modifying therapy since the end of the base study and planning to continue taking a statin throughout the study

Exclusion Criteria:

* History of heart failure, arrhythmias, heart attack, unstable angina, or stroke within 3 months prior to screening, uncontrolled blood pressure, uncontrolled high cholesterol or liver disease.
* History of mental instability, drug/alcohol abuse within the past 5 years
* Pregnant or breast-feeding
* History of cancer within the last 5 years
* HIV positive
* Donated blood products within 8 weeks
* Currently participating or have participated in a study with an investigational compound within the last 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1623 (Actual)
Dates: Start 2008-03-24 (Actual); Primary Completion 2009-07-02 (Actual); Study Completion 2017-11-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Low Density Lipoprotein Cholesterol | Baseline and 24 weeks
Number of participants with hepatitis-related adverse experiences | Through 88 weeks
Number of participants with Alanine Transaminase consecutive elevations greater than or equal to 3xULN (Upper Limit of Normal) | Through 88 weeks
Number of participants with Aspartate Aminotransferase consecutive elevations greater than or equal to 3xULN | Through 88 weeks
Number of participants with Creatine Phosphokinase elevations greater than or equal to 10xULN | Through 88 weeks
Number of participants with Creatine Phosphokinase elevations greater than or equal 10xULN with muscle symptoms | Through 88 weeks
Number of participants with sodium, chloride, or bicarbonate elevations greater than ULN | Through 88 weeks
Number of participants with reduction in potassium levels less than LLN (Lower Limit of Normal) | Through 88 weeks
Number of participants with myalgia | Through 88 weeks
Number of participants with rhabdomyolysis | Through 88 weeks
Number of participants with pre-specified adjudicated cardiovascular serious adverse events | Through 88 weeks
Number of participants with death from any cause | Through 88 weeks
Number of participants with significant increase in Blood Pressure | Through 88 weeks

SECONDARY OUTCOMES:
Change from baseline in High Density Lipoprotein Cholesterol | Baseline, 24 weeks, and 76 weeks
Change from baseline in non-High Density Lipoprotein Cholesterol | Baseline, 24 weeks, and 76 weeks
Change from baseline in Apolipoprotein B | Baseline, 24 weeks, and 76 weeks
Change from baseline in Apolipoprotein A-1 | Baseline, 24 weeks, and 76 weeks
Change from baseline in Low Density Lipoprotein Cholesterol | Baseline, 24 weeks, and 76 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] Brinton EA, Kher U, Shah S, Cannon CP, Davidson M, Gotto AM, Ashraf TB, McCrary Sisk C, Dansky H, Mitchel Y, Barter P; DEFINE Investigators. Effects of anacetrapib on plasma lipids in specific patient subgroups in the DEFINE (Determining the Efficacy and Tolerability of CETP INhibition with AnacEtrapib) trial. J Clin Lipidol. 2015 Jan-Feb;9(1):65-71. doi: 10.1016/j.jacl.2014.10.005. Epub 2014 Nov 4. PMID 25670362
- [Derived] Gotto AM Jr, Kher U, Chatterjee MS, Liu Y, Li XS, Vaidya S, Cannon CP, Brinton EA, Moon JE, Shah S, Dansky HM, Mitchel Y, Barter P; DEFINE Investigators. Lipids, safety parameters, and drug concentrations after an additional 2 years of treatment with anacetrapib in the DEFINE study. J Cardiovasc Pharmacol Ther. 2014 Nov;19(6):543-9. doi: 10.1177/1074248414529621. Epub 2014 Apr 14. PMID 24737712
- [Derived] Cannon CP, Shah S, Dansky HM, Davidson M, Brinton EA, Gotto AM, Stepanavage M, Liu SX, Gibbons P, Ashraf TB, Zafarino J, Mitchel Y, Barter P; Determining the Efficacy and Tolerability Investigators. Safety of anacetrapib in patients with or at high risk for coronary heart disease. N Engl J Med. 2010 Dec 16;363(25):2406-15. doi: 10.1056/NEJMoa1009744. Epub 2010 Nov 17. PMID 21082868
- [Derived] Cannon CP, Dansky HM, Davidson M, Gotto AM Jr, Brinton EA, Gould AL, Stepanavage M, Liu SX, Shah S, Rubino J, Gibbons P, Hermanowski-Vosatka A, Binkowitz B, Mitchel Y, Barter P; DEFINE investigators. Design of the DEFINE trial: determining the EFficacy and tolerability of CETP INhibition with AnacEtrapib. Am Heart J. 2009 Oct;158(4):513-519.e3. doi: 10.1016/j.ahj.2009.07.028. PMID 19781408